CLINICAL TRIAL: NCT02328599
Title: A Prospective Consortium Evaluating the Long-term Follow-up of Patients With Type 2 Diabetes Enrolled In a Randomized Controlled Trial Comparing Bariatric Surgery Versus Medical Management
Brief Title: Alliance of Randomized Trials of Medicine vs Metabolic Surgery in Type 2 Diabetes
Acronym: ARMMS-T2D
Status: Enrolling by invitation | Type: Observational
Sponsor: Ali Aminian (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Ali Aminian, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: COV EES-14606; U01DK114156 (NIH)
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Study specific blood and urine specimens will be analyzed at a central laboratory. Participation in the research repository is optional. Blood will be drawn and stored at each site for later analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical: Prior Bariatric surgery
  Interventions: Procedure: Bariatric surgery involving Roux-en-Y gastric bypass; Procedure: Bariatric surgery involving Laparoscopic adjustable gastric banding; Procedure: Bariatric surgery involving Laparoscopic sleeve gastrectomy
- Non-surgical: Medical / Lifestyle management

INTERVENTIONS:
Procedure: Bariatric surgery involving Roux-en-Y gastric bypass — Subjects previously underwent Bariatric surgery involving Roux-en-Y gastric bypass (RYGB) surgery at one of the 4 participating sites and will be followed prospectively.
  Other Names: RYGB
  Groups: Surgical
Procedure: Bariatric surgery involving Laparoscopic adjustable gastric banding — Subjects previously underwent Bariatric surgery involving laparoscopic adjustable gastric banding (LAGB) surgery at one of the 4 participating sites and will be followed prospectively.
  Other Names: LAGB
  Groups: Surgical
Procedure: Bariatric surgery involving Laparoscopic sleeve gastrectomy — Subjects previously underwent Bariatric surgery involving laparoscopic sleeve gastrectomy (LSG) surgery at one of the 4 participating sites and will be followed prospectively.
  Other Names: LSG
  Groups: Surgical

SUMMARY:
Initially, 4 teams of investigators conducted randomized controlled trials (RCT) at their own site to evaluate the effectiveness of bariatric surgery compared to medical/lifestyle management of type 2 diabetes. Each study followed subjects for a duration of about 1 - 3 years. Following this, a consortium was created to pool data and continue to follow study participants. This early collaboration of the 4 groups of investigators was supported by Industry sponsors (Ethicon, Inc and Medtronic-MITG). Now, the investigators have successfully received a grant from the NIH, as the sole supporter of continued observational follow-up of study participants.

The continuing aim of this study is to combine data from the 4 studies and follow the original randomized subjects for an additional 5 years of follow-up. The purpose of the study is to determine the longer term durability and effectiveness of bariatric surgery compared to medical/lifestyle intervention on the treatment of type 2 diabetes.

DETAILED DESCRIPTION:
The four investigative groups initiated their individual RCT's at their respective sites to evaluate the effectiveness of bariatric surgery compared to multidisciplinary medical and lifestyle management of diabetes and body weight. The original trials were each designed to assess feasibility over a relatively short duration of follow-up (1-3 years). Individually, each trial lacked the sample size and duration of follow-up to meaningfully inform clinical decision making. Together, with the funding provided by the NIH for longer follow-up, the Consortium trial can provide a unique national resource to address timely and unanswered clinical questions related to the durability of these alternative management approaches in patients with T2D and obesity. Together, participants from these studies represent the largest cohort with diabetes (one third having a BMI <35 kg/m2) ever to undergo randomized assignment to bariatric surgical procedure vs. medical/lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

* Original inclusion criteria for participation in the RCTs at all sites included:

  * Candidate for general anesthesia or unsupervised exercise.
  * Age ≥20 and ≤65 years.
  * Body mass index >27 and ≤45 kg/m2.
  * Diagnosis of type 2 diabetes confirmed by either requiring diabetes medication and/or having elevated glycemia based on HbA1c, fasting plasma glucose, and/or oral glucose tolerance test (OGTT) results, according to American Diabetes Association criteria.
  * Ability and willingness to participate in the study and agree to any of the research arms.
  * Able to understand the options and to comply with the requirements of each program.
  * Negative urine pregnancy test at screening and baseline visits (prior to surgery) for women of childbearing potential (i.e., biologically capable of becoming pregnant).

Exclusion Criteria:

* Subjects who were randomized in one of the four RCTs but never initiated intervention / did not receive randomized treatment
* Refusal to sign informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who were previously enrolled in a Randomized Control Trial (RCT) at one of the four participating sites who initiated one of the intervention procedures - bariatric surgery or medical/lifestyle therapy.
Sampling Method: Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 7 years and up to 13 years for earliest enrollees
  Between group (medical vs. surgical) in HbA1c from baseline to 7 year for all participants and up to 13 years for the earliest enrollees

SECONDARY OUTCOMES:
HbA1c < 6.5% | 7 years and each annual visit through the last known follow-up for all patients up to 13 years
  percent of those achieving diabetes remission without the need for anti-diabetic medications

OTHER OUTCOMES:
HbA1c >6.5% | 7-13 years
  relapse in diabetes control requiring the addition of anti-diabetic medications
change in body weight measured in BMI | 7 years and up to 13 years for earliest enrollees
  Change in body weight status from baseline
change in fasting glucose | 7 years and up to 13 years for earliest enrollees
  Change in diabetes related outcomes including cardiovascular risk factors
change in cholesterol levels | 7 years and up to 13 years for earliest enrollees
  Change in diabetes related outcomes including cardiovascular risk factors
change in blood pressure | 7 years and up to 13 years for earliest enrollees
  Change in diabetes related outcomes including cardiovascular risk factors
change in albuminuria | 7 years and up to 13 years for earliest enrollees
  Change in diabetes related outcomes including cardiovascular risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Aminian Ali, MD, Principal Investigator — The Cleveland Clinic; John Kirwan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (4):
- United States (4):
  - Joslin Diabetes Center, Boston, Massachusetts
  - Cleveland Clinic Digestive Disease Institute, Cleveland, Ohio
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] Carlsson LM, Peltonen M, Ahlin S, Anveden A, Bouchard C, Carlsson B, Jacobson P, Lonroth H, Maglio C, Naslund I, Pirazzi C, Romeo S, Sjoholm K, Sjostrom E, Wedel H, Svensson PA, Sjostrom L. Bariatric surgery and prevention of type 2 diabetes in Swedish obese subjects. N Engl J Med. 2012 Aug 23;367(8):695-704. doi: 10.1056/NEJMoa1112082. PMID 22913680
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Schauer PR, Burguera B, Ikramuddin S, Cottam D, Gourash W, Hamad G, Eid GM, Mattar S, Ramanathan R, Barinas-Mitchel E, Rao RH, Kuller L, Kelley D. Effect of laparoscopic Roux-en Y gastric bypass on type 2 diabetes mellitus. Ann Surg. 2003 Oct;238(4):467-84; discussion 84-5. doi: 10.1097/01.sla.0000089851.41115.1b. PMID 14530719
- [Background] Rubino F, Schauer PR, Kaplan LM, Cummings DE. Metabolic surgery to treat type 2 diabetes: clinical outcomes and mechanisms of action. Annu Rev Med. 2010;61:393-411. doi: 10.1146/annurev.med.051308.105148. PMID 20059345
- [Background] Brethauer SA, Aminian A, Romero-Talamas H, Batayyah E, Mackey J, Kennedy L, Kashyap SR, Kirwan JP, Rogula T, Kroh M, Chand B, Schauer PR. Can diabetes be surgically cured? Long-term metabolic effects of bariatric surgery in obese patients with type 2 diabetes mellitus. Ann Surg. 2013 Oct;258(4):628-36; discussion 636-7. doi: 10.1097/SLA.0b013e3182a5034b. PMID 24018646
- [Background] Dixon JB, O'Brien PE, Playfair J, Chapman L, Schachter LM, Skinner S, Proietto J, Bailey M, Anderson M. Adjustable gastric banding and conventional therapy for type 2 diabetes: a randomized controlled trial. JAMA. 2008 Jan 23;299(3):316-23. doi: 10.1001/jama.299.3.316. PMID 18212316
- [Background] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Background] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317
- [Background] Ikramuddin S, Korner J, Lee WJ, Connett JE, Inabnet WB, Billington CJ, Thomas AJ, Leslie DB, Chong K, Jeffery RW, Ahmed L, Vella A, Chuang LM, Bessler M, Sarr MG, Swain JM, Laqua P, Jensen MD, Bantle JP. Roux-en-Y gastric bypass vs intensive medical management for the control of type 2 diabetes, hypertension, and hyperlipidemia: the Diabetes Surgery Study randomized clinical trial. JAMA. 2013 Jun 5;309(21):2240-9. doi: 10.1001/jama.2013.5835. PMID 23736733
- [Background] Halperin F, Ding SA, Simonson DC, Panosian J, Goebel-Fabbri A, Wewalka M, Hamdy O, Abrahamson M, Clancy K, Foster K, Lautz D, Vernon A, Goldfine AB. Roux-en-Y gastric bypass surgery or lifestyle with intensive medical management in patients with type 2 diabetes: feasibility and 1-year results of a randomized clinical trial. JAMA Surg. 2014 Jul;149(7):716-26. doi: 10.1001/jamasurg.2014.514. PMID 24899464
- [Background] Courcoulas AP, Goodpaster BH, Eagleton JK, Belle SH, Kalarchian MA, Lang W, Toledo FG, Jakicic JM. Surgical vs medical treatments for type 2 diabetes mellitus: a randomized clinical trial. JAMA Surg. 2014 Jul;149(7):707-15. doi: 10.1001/jamasurg.2014.467. PMID 24899268
- [Background] Arterburn DE, Bogart A, Sherwood NE, Sidney S, Coleman KJ, Haneuse S, O'Connor PJ, Theis MK, Campos GM, McCulloch D, Selby J. A multisite study of long-term remission and relapse of type 2 diabetes mellitus following gastric bypass. Obes Surg. 2013 Jan;23(1):93-102. doi: 10.1007/s11695-012-0802-1. PMID 23161525
- [Background] Cummings DE, Flum DR. Gastrointestinal surgery as a treatment for diabetes. JAMA. 2008 Jan 23;299(3):341-3. doi: 10.1001/jama.299.3.341. No abstract available. PMID 18212321
- [Background] Rubino F, Forgione A, Cummings DE, Vix M, Gnuli D, Mingrone G, Castagneto M, Marescaux J. The mechanism of diabetes control after gastrointestinal bypass surgery reveals a role of the proximal small intestine in the pathophysiology of type 2 diabetes. Ann Surg. 2006 Nov;244(5):741-9. doi: 10.1097/01.sla.0000224726.61448.1b. PMID 17060767
- [Background] Zimmet P, Alberti KG, Rubino F, Dixon JB. IDF's view of bariatric surgery in type 2 diabetes. Lancet. 2011 Jul 9;378(9786):108-10. doi: 10.1016/S0140-6736(11)61027-1. No abstract available. PMID 21742162
- [Background] Sjostrom L, Peltonen M, Jacobson P, Sjostrom CD, Karason K, Wedel H, Ahlin S, Anveden A, Bengtsson C, Bergmark G, Bouchard C, Carlsson B, Dahlgren S, Karlsson J, Lindroos AK, Lonroth H, Narbro K, Naslund I, Olbers T, Svensson PA, Carlsson LM. Bariatric surgery and long-term cardiovascular events. JAMA. 2012 Jan 4;307(1):56-65. doi: 10.1001/jama.2011.1914. PMID 22215166
- [Background] Longitudinal Assessment of Bariatric Surgery (LABS) Consortium; Flum DR, Belle SH, King WC, Wahed AS, Berk P, Chapman W, Pories W, Courcoulas A, McCloskey C, Mitchell J, Patterson E, Pomp A, Staten MA, Yanovski SZ, Thirlby R, Wolfe B. Perioperative safety in the longitudinal assessment of bariatric surgery. N Engl J Med. 2009 Jul 30;361(5):445-54. doi: 10.1056/NEJMoa0901836. PMID 19641201
- [Background] Adams TD, Davidson LE, Litwin SE, Kolotkin RL, LaMonte MJ, Pendleton RC, Strong MB, Vinik R, Wanner NA, Hopkins PN, Gress RE, Walker JM, Cloward TV, Nuttall RT, Hammoud A, Greenwood JL, Crosby RD, McKinlay R, Simper SC, Smith SC, Hunt SC. Health benefits of gastric bypass surgery after 6 years. JAMA. 2012 Sep 19;308(11):1122-31. doi: 10.1001/2012.jama.11164. PMID 22990271
- [Background] Rubino F, Kaplan LM, Schauer PR, Cummings DE; Diabetes Surgery Summit Delegates. The Diabetes Surgery Summit consensus conference: recommendations for the evaluation and use of gastrointestinal surgery to treat type 2 diabetes mellitus. Ann Surg. 2010 Mar;251(3):399-405. doi: 10.1097/SLA.0b013e3181be34e7. PMID 19934752
- [Background] O'Brien PE, Dixon JB, Laurie C, Skinner S, Proietto J, McNeil J, Strauss B, Marks S, Schachter L, Chapman L, Anderson M. Treatment of mild to moderate obesity with laparoscopic adjustable gastric banding or an intensive medical program: a randomized trial. Ann Intern Med. 2006 May 2;144(9):625-33. doi: 10.7326/0003-4819-144-9-200605020-00005. PMID 16670131
- [Background] Maggard-Gibbons M, Maglione M, Livhits M, Ewing B, Maher AR, Hu J, Li Z, Shekelle PG. Bariatric surgery for weight loss and glycemic control in nonmorbidly obese adults with diabetes: a systematic review. JAMA. 2013 Jun 5;309(21):2250-61. doi: 10.1001/jama.2013.4851. PMID 23736734
- [Background] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Brethauer SA, Navaneethan SD, Aminian A, Pothier CE, Kim ES, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric surgery versus intensive medical therapy for diabetes--3-year outcomes. N Engl J Med. 2014 May 22;370(21):2002-13. doi: 10.1056/NEJMoa1401329. Epub 2014 Mar 31. PMID 24679060
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] CDC. National Diabetes Statistics Report: Estimates of Diabetes and Its Burden in the United States, 2014. US Department of Health and Human Services.
- [Derived] Patti ME, Hu B, Kirschling S, Wang HJ, Foster K, Sarig Y, Simonson DC, Wolfs D, Arterburn D, O'Brien MJ, Vernon AH, Jakicic JM, Laffel L, Ojukwu S, Kashyap SR, Aminian A, Schauer PR, Cummings DE, Gourash WF, Courcoulas A, Kirwan JP. Effect of Social Vulnerability on Efficacy of Bariatric Surgery Versus Medical and Lifestyle Intervention for Type 2 Diabetes: Analysis of the ARMMS-T2D Consortium of Randomized Trials. Ann Intern Med. 2026 Jan 20. doi: 10.7326/ANNALS-24-01882. Online ahead of print. PMID 41554124
- [Derived] Courcoulas AP, Patti ME, Hu B, Arterburn DE, Simonson DC, Gourash WF, Jakicic JM, Vernon AH, Beck GJ, Schauer PR, Kashyap SR, Aminian A, Cummings DE, Kirwan JP. Long-Term Outcomes of Medical Management vs Bariatric Surgery in Type 2 Diabetes. JAMA. 2024 Feb 27;331(8):654-664. doi: 10.1001/jama.2024.0318. PMID 38411644
- [Derived] Kirwan JP, Courcoulas AP, Cummings DE, Goldfine AB, Kashyap SR, Simonson DC, Arterburn DE, Gourash WF, Vernon AH, Jakicic JM, Patti ME, Wolski K, Schauer PR. Diabetes Remission in the Alliance of Randomized Trials of Medicine Versus Metabolic Surgery in Type 2 Diabetes (ARMMS-T2D). Diabetes Care. 2022 Jul 7;45(7):1574-1583. doi: 10.2337/dc21-2441. PMID 35320365